CLINICAL TRIAL: NCT02332577
Title: A Multi-centre, Non-inferiority, Randomized, Double-blind, Phase IV Study Comparing Pristinamycin (2g x 2 Per Day for 2 Days Then 1g x 3 Per Day for 5 to 7 Days) to Amoxicillin (1g x 3 Per Day) for 7 to 9 Days in Adults With Acute Community Acquired Pneumonia With a PORT Score of II or III
Brief Title: Study to Compare the Efficacy of Pristinamycin (Pyostacine ®) Versus Amoxicillin in the Treatment of Acute Community Acquired Pneumonia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor stopped the study due to low recruitment with no safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRISTL06562; U1111-1160-6001 (Other: UTN)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Pristinamycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pristinamycin + Placebo (Experimental): Pristinamycin: 500 mg tablet, 4 tablets x 2/day for 2 days then 2 tablets x 3/day for 5 to 7 days Amoxicillin Placebo: capsule, 2 capsules x 3 /day for 7 to 9 days.
  Interventions: Drug: PRISTINAMYCIN XRP7263; Drug: Amoxicillin Placebo
- Amoxicillin + Placebo (Active Comparator): Amoxicillin: 500 mg capsule, 2 capsules x 3/day for 7 to 9 days Pristinamycin Placebo: tablet, 4 tablets x 2/day for 2 days then 2 tablets x 3/day for 5 to 7 days.
  Interventions: Drug: Amoxicillin; Drug: PRISTINAMYCIN Placebo

INTERVENTIONS:
Drug: PRISTINAMYCIN XRP7263 — Pharmaceutical form:tablet 500 mg Route of administration: oral
  Other Names: Pyostacine ®
  Arms: Pristinamycin + Placebo
Drug: Amoxicillin — Pharmaceutical form:capsule 500 mg Route of administration: oral
  Other Names: Amoxicilline EG
  Arms: Amoxicillin + Placebo
Drug: Amoxicillin Placebo — Pharmaceutical form: capsule Route of administration: oral
  Arms: Pristinamycin + Placebo
Drug: PRISTINAMYCIN Placebo — Pharmaceutical form:Tablet Route of administration: Oral
  Arms: Amoxicillin + Placebo

SUMMARY:
Primary Objective:

To evaluate the clinical efficacy of pristinamycin at a dose of 2g x 2/day for 2 days then 1g x 3/day for 5 to 7 days versus amoxicillin 1g x3 /day for 7 to 9 days, 5 to 9 days after the end of treatment.

Secondary Objectives:

To evaluate the clinical efficacy in a subpopulation bacteriologically documented at inclusion and according to procalcitonin level.

To evaluate the efficacy of treatments against pneumococcus. To evaluate the rate of relapse and mortality 30±2 days after treatment is started.

To document failures. To collect and follow up adverse events.

DETAILED DESCRIPTION:
The total study duration for each patient is 1 month with a treatment period of 7 to 9 days and a follow-up period of 21 to 23 days.

ELIGIBILITY:
Inclusion criteria:

Male or female more than 18 years old with a presumed bacterial acute community acquired pneumonia presenting a PORT score of II or III (Fine II or III).

The acute community acquired pneumonia is defined by:

* Pulmonary x-ray (carried out within the 48 hours prior to randomization) showing new lobar or multilobar infiltrates.
* At least 4 functional and/or clinical symptoms from among the following:
* Fever characterized by a temperature of more than 38.5 at least once within 24h prior to inclusion.
* Appearance or aggravation of a cough.
* Appearance of purulent expectoration.
* Appearance or aggravation of dyspnoea.
* Tachypnoea
* Chest pain
* A characteristic sign on percussion and/or auscultation associated with a pulmonary condensation focus.

Exclusion criteria:

Patients having been diagnosed with legionellosis.

Patients having received systemic antibiotic therapy of over 24 hours within the week preceding the start of study treatment.

Associated neoplasm (active cancer [of whatever type, solid or haematological] or diagnosed within the year other than basocellular skin cancer).

Severe or very severe chronic obstructive pulmonary disease (COPD) (GOLD3 and GOLD4).

History of bacterial pneumonia in the past 12 months.

Bronchopulmonary diseases likely to interfere with the assessment of the therapeutic response.

Known hypersensitivity to streptogramins, penicillin and other betalactamines or excipients of the treatments studied.

History of severe skin reaction after taking pristinamycin or amoxicillin.

Kidney disease (chronic kidney failure or creatinine clearance ≤30 mL/minute).

Patients treated with allopurinol, colchicine, immunosuppressants (cyclosporin, tacrolimus, mycophenolate mofetil, methotrexate, biotherapies) oral anticoagulants in the previous 6 months or during the study.

Known HIV infection, whatever the stage.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients cured established from the clinical course and pulmonary radiological course | 5 to 9 days post-treatment

SECONDARY OUTCOMES:
Percentage of cured patients evaluated by bacteriological documentation and procalcitonin levels | 5 to 9 days post-treatment
Percentage of cured patients evaluated by bacteriological documentation for pneumococcus | 5 to 9 days post-treatment
Percentage of patients with relapse | at Day 30
Mortality rate | at Day 30
Number of documented failures | 5 to 9 days post-treatment
Proportion of patients with adverse events | up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- France (11):
  - Investigational Site Number :250029, Avoine
  - Investigational Site Number :250015, Colombes
  - Investigational Site Number :250010, Grenoble
  - Investigational Site Number :250032, La Riche
  - Investigational Site Number :250054, Monaco Cedex
  - Investigational Site Number :250023, Nantes
  - Investigational Site Number :250022, Paris
  - Investigational Site Number :250004, Pringy
  - Investigational Site Number :250001, Saint-Priest-en-Jarez
  - Investigational Site Number :250031, Segré
  - Investigational Site Number :250034, Tours
- Tunisia (8):
  - Investigational Site Number :788001, Aryanah
  - Investigational Site Number :788002, Aryanah
  - Investigational Site Number :788004, Aryanah
  - Investigational Site Number :788005, Aryanah
  - Investigational Site Number :788014, La Marsa
  - Investigational Site Number :788007, Monastir
  - Investigational Site Number :788011, Monastir
  - Investigational Site Number :788009, Sfax

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org